CLINICAL TRIAL: NCT02707809
Title: Effects of Perioperative Dexmedetomidine Infusion on Microcirculation and Kidney and Intestinal Injury in Kidney Transplant Recipients
Brief Title: Effects of Dexmedetomidine on Microcirculation of Kidney Transplant Recipient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201512039MINB
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-04

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Routine anesthesia care for kidney transplant
- Dexmedetomidine (Experimental): Routine anesthesia care for kidney transplant and perioperative intravenous infusion of dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
The microcirculation is altered in acute kidney injury and chronic kidney disease. The microcirculation is poor in end-stage renal disease patients receiving hemodialysis. Kidney transplant can improve the life quality of these patients. However, surgical stress and inflammatory response may cause microcirculatory dysfunction and intestinal injury. Moreover, the transplanted kidney would suffer from the ischemia and reperfusion injury, and it may result in acute kidney injury. In ischemia and reperfusion injury animal model, dexmedetomidine has been proven to attenuate kidney and intestinal injury. In our previous study of surgical stress and pain stimulation rat model, we found that dexmedetomidine attenuate the intestinal microcirculatory dysfunction. In patients receiving coronary artery bypass graft surgery, dexmedetomidine increases urine output and decreases postoperative serum level of neutrophil gelatinase-associated lipocalin.

This study aims to investigate whether perioperative dexmedetomidine infusion may attenuate microcirculatory dysfunction, kidney injury, and intestinal injury for patients undergoing kidney transplant.

DETAILED DESCRIPTION:
The microcirculation is altered in acute kidney injury and chronic kidney disease. The microcirculation is poor in end-stage renal disease patients receiving hemodialysis. Kidney transplant can improve the life quality of these patients. However, surgical stress and inflammatory response may cause microcirculatory dysfunction and intestinal injury. Moreover, the transplanted kidney would suffer from the ischemia and reperfusion injury, and it may result in acute kidney injury. In ischemia and reperfusion injury animal model, dexmedetomidine has been proven to attenuate kidney and intestinal injury. In our previous study of surgical stress and pain stimulation rat model, we found that dexmedetomidine attenuate the intestinal microcirculatory dysfunction. In patients receiving coronary artery bypass graft surgery, dexmedetomidine increases urine output and decreases postoperative serum level of neutrophil gelatinase-associated lipocalin. The aim of this study is to investigate whether perioperative dexmedetomidine infusion may attenuate microcirculatory dysfunction, kidney injury, and intestinal injury for patients undergoing kidney transplant.

This is a randomized, single-blind, prospective, controlled clinical trial. The patients will be randomly assigned to the control group or dexmedetomidine group. After induction of anesthesia, the patients in the control group will receive regular perioperative care. The patients in the dexmedetomidine group will receive perioperative dexmedetomidine continuous intravenous infusion after induction of anesthesia till 2 hours after the end of the operation. All patients will receive sublingual microcirculation examination, laboratory tests of blood urine nitrogen, creatinine, and enzyme-linked immunosorbent assays of serum level of endocan, diamine oxidase, and neutrophil gelatinase-associated lipocalin at preset time points. The urine level of neutrophil gelatinase-associated lipocalin will also be measured. The vital signs and urine output will be recorded. The difference between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipient

Exclusion Criteria:

* allergic history to dexmedetomidine
* refractory bradycardia < 60 bpm despite treatment
* severe atrioventricular block (2nd and 3rd degree)
* previous operation of tongue

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Total small vessel density of sublingual microcirculation | Postoperative 2h
  Sublingual microcirculation captured using an incident dark-field video microscope
Creatinine level | Postoperative day 2
  Difference in serum creatine levels between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No